CLINICAL TRIAL: NCT01237886
Title: Weaning And Variability Evaluation
Acronym: WAVE
Status: Completed | Type: Observational
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2009-569
Record Dates: First submitted 2010-10-13; First posted 2010-11-10 (Estimated); Last update posted 2017-07-07 (Actual); Status verified 2017-07

CONDITIONS: Mechanically Ventilated Patients; Extubation
Keywords: spontaneous breathing trial; heart rate variability; respiratory rate variability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Knowing when to liberate patients from mechanical ventilation (i.e. removal of breathing or endotracheal tube or extubation) is critically important, as both prolonged ventilation and failed extubation are both associated with harm and risk of death. Our objective is to improve the safety of extubation by harnessing hidden information contained in the patterns of variation of heart and respiratory rate measured over intervals-in-time. Currently, to assess a patient's ability to be extubated, a spontaneous breathing trial (SBT) is routinely performed, where the level of ventilator support is reduced, and their response is observed in order to help predict if they will tolerate extubation (i.e. complete removal of ventilator support). Given that health is associated with a high degree of variation of physiologic parameters (e.g. heart and respiratory rate), and illness & stress are associated with a loss of variability, the investigators aim to uncover the loss of variation as a measure of stress during SBT's. The investigators hypothesize that maintaining stable heart rate and respiratory rate variability (HRV and RRV) throughout the SBT will predict subsequent successful extubation, and conversely, a reduction in either HRV or RRV manifest during a SBT predicts extubation failure. A pilot study has demonstrated feasibility, and compelling preliminary results. A website, centralized data storage and analysis, and a trans-disciplinary team of scientists are in place to definitively test this novel technology. Determination of when to extubate critically ill patients remains a high-stakes clinical challenge; and improved prediction of extubation failure has potential to save lives and reduce costs in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Invasive mechanical ventilation for >48 hours,
* patient is ready for SBTs for assessment for extubation,
* has a normal sinus rhythm at time of SBT (no pacemaker),
* is tolerating pressure support ventilation ≤14 cm H2O (SpO2 ≥ 90% with FiO2 ≤ 40% and PEEP ≤ 10 cm H2O),
* hemodynamically stable (low or no vasopressors), stable neurological status (no deterioration in GCS during prior 24 hours & ICP < 20),
* intact airway reflexes (cough & gag).

Exclusion Criteria:

* Order not to re-intubate,
* anticipated withdrawal of life support,
* known or suspected severe weakness (myopathy, neuropathy or quadriplegia),
* tracheostomy,
* and prior extubation during ICU stay.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ICU patients
Sampling Method: Non-Probability Sample
Enrollment: 660 (Actual)
Dates: Start 2009-11; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Continuous heart rate (electrocardiogram) & respiratory rate (CO2 capnography) waveforms | at time of spontaneous breathing trial (at least 48 hours after intubation and within 24 hours of extubation)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Seely, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (14):
- United States (7):
  - The University of Michigan Medical Center, Ann Arbor, Michigan
  - Billings Clinic, Billings, Montana
  - Dartmouth Hitchcock Memorial Hospital, Lebanon, New Hampshire
  - Columbia University, New York, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Intermountain Medical Center/University of Utah School of Medicine, Salt Lake City, Utah
- Canada (7):
  - The University of British Columbia, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - The Ottawa Hospital-Civic Campus, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Mt Sinai, Toronto, Ontario

REFERENCES:
- [Derived] Seely AJ, Bravi A, Herry C, Green G, Longtin A, Ramsay T, Fergusson D, McIntyre L, Kubelik D, Maziak DE, Ferguson N, Brown SM, Mehta S, Martin C, Rubenfeld G, Jacono FJ, Clifford G, Fazekas A, Marshall J; Canadian Critical Care Trials Group (CCCTG). Do heart and respiratory rate variability improve prediction of extubation outcomes in critically ill patients? Crit Care. 2014 Apr 8;18(2):R65. doi: 10.1186/cc13822. PMID 24713049